CLINICAL TRIAL: NCT06804499
Title: Tampere Coronary Artery Disease and Sudden Cardiac Arrest Study
Acronym: CADSCA
Status: Recruiting | Type: Observational
Sponsor: Tampere Heart Hospital (Other)
Collaborators: Tampere University (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Jussi Hernesniemi, Research Director, Tampere University Hospital
Other Study IDs: R24037
Record Dates: First submitted 2025-01-14; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Sudden Cardiac Arrest; Sudden Cardiac Death; Sudden Cardiac Death Due to Cardiac Arrhythmia; Coronary Arterial Disease (CAD); Acute Coronary Event
Keywords: sudden cardiac death; sudden cardiac arrest; coronary artery disease; acute coronary syndrome
MeSH Terms: conditions — Death, Sudden, Cardiac; Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Coronary Artery Disease: The study will recruit adult patients diagnosed with coronary artery disease (CAD) who are living in the Wellbeing Services County of Pirkanmaa. CAD must be with an invasive coronary angiogram or computed tomography angiogram (CTA), which cardiologists evaluate based on current guidelines for stenosis level evaluation and fractional flow reserve (FFR) results. An invasive coronary angiogram or CTA must be done within three (3) months before recruitment. The study subjects must have a good or moderate everyday functional ability.
  The study is non-interventional.

SUMMARY:
The goal of this observational study is to recognize clinical and genetic risk factors for sudden cardiac arrest (SCA) and death (SCD) in patients with coronary artery disease (CAD).

The main questions it aims to answer are:

Are we able to recognize clinical or treatment-related risk factors for SCA or SCD? Can we identify new genetic risk factors for SCA or SCD in patients under 75 years?

Participants diagnosed with CAD answer a short survey about their medical history and socioeconomic status. A standard ECG addition to a five (5) minute ECG recording is taken from all the study subjects. In addition to a few short physiological tests (e.g. blood pressure, height, weight, grip strength), a blood sample is withdrawn from a selected group of study subjects.

Medical healthcare records are used to follow all study subjects, and no follow-up visits are required.

DETAILED DESCRIPTION:
Source data verification is not planned for the baseline data acquisition. SCD data is collected from the national death certificate register, which is mandated by Finnish legislation. Death certificates must include information about all the significant prevalent diseases and the events and circumstances leading to death. Also, data regarding the cause of death (ICD-10 classification) and the place of death must be included. The certificate is written by the last physician treating the patient and is complemented with medical or medicolegal autopsy results if available. Research members will fully review all detected SCD case from medical records and death certificates.

Patients treated for CAD in Tampere Heart Hospital are recruited by research staff according to up-to-date Standard Operating Procedures (SOP). Research staff will conduct surveys and physiological measurements and take a blood sample in as planned. The blood sample is processed and stored according to research plan. The collected data is entered and saved to the Tampere Heart Hospital RedCap database. All research staff is trained according to up-to-date SOP. The final analytics of the blood samples including genetic testing will be decided later.

The study is designed to have 80% power (alpha 0.05) to demonstrate a small-medium effect (Cohen's D 0.2-0.5) for normally distributed variables. To this end, 150-200 SCD cases should be detected in the follow-up. Based on previous research, 4000 subjects with four years of follow-up need to be recruited to fulfil the target number of SCD cases. With this sample, a 2.5-3.5 times risk ratio for categorical variables could be detected (80% power).

Missing data will be addressed as such. If significant number of study subjects with missing data will be detected data imputing can be considered during analysis.

Prospective data regarding SCD will be analyzed in addition to conventional statistical methods, with Cox regression model. Also Fine Gray subdistribution models will be used. Machine learning model can used especially analyzing ECG and genetic data.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. A patient who lives in the area of 'Wellbeing Services County of Pirkanmaa' and seeks treatment for coronary artery disease (CAD).
3. CAD is diagnosed with invasive coronary angiogram or computed tomography angiogram (CTA) which is evaluated by cardiologists based on current guidelines for stenosis level evaluation and fractional flow reserve (FFR) results.
4. An invasive coronary angiogram or CTA is done within three (3) months.
5. Good or moderate everyday functional ability

Exclusion Criteria:

1. Life expectancy <1 months.
2. A significant valvular heart disease treated previously (endovascular or surgical) or requires treatment (endovascular or surgical) in the next three (3) months.
3. Previously implanted cardioverter-defibrillators (ICD) or will be implanted in the next three (3) months.
4. An active malignancy (ongoing treatment for a solid tumour, metastatic solid tumour, fast progressing haematological malignancy, or equal malignant disease).
5. A significant neurodegenerative disease (dementia, Mini-Mental State Examination (MMSE) <23 or equivalenneurodegenerative disease affecting everyday functional ability, like ALS, myositis, prograded MS-disease or Parkinson's disease).
6. Intellectual disability or a significant disability affecting cognitive functions
7. Do-not-resuscitate (DNR) treatment decision

Subgroup with blood samples:

Blood samples are withdrawn from all study subjects under 76 years of age. Additionally, PaxGene samples are withdrawn from i) all study subjects under 65 years of age and ii) subjects between 65-76 years, if they have detected QRS-time>110ms in the latest ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit adult patients diagnosed with coronary artery disease (CAD) who are living in the Wellbeing Services County of Pirkanmaa. CAD must be with an invasive coronary angiogram or computed tomography angiogram (CTA), which cardiologists evaluate based on current guidelines for stenosis level evaluation and fractional flow reserve (FFR) results. An invasive coronary angiogram or CTA must be done within three (3) months before recruitment. The study subjects must have a good or moderate everyday functional ability.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
Sudden Cardiac Death (SCD) | 15 years
  The primary endpoints of the study are sudden cardiac death (SCD) and sudden cardiac arrest (SCA).
  A SCD is defined as:
  * a cardiac death within one hour from the beginning of symptoms,
  * or if the patient is found dead (cardiac causes) but is known to have a good clinical condition within 24 hours and
  A SCA is defined as:
  * a hemodynamical collapse by cardiac cause and not influenced by trauma, drowning, respiratory insufficiency, drug overdose, or other non-cardiac cause.
  * There are no limitations on symptom duration.

SECONDARY OUTCOMES:
Secondary endpoints | 15 years
  Secondary endpoint include significant cardiovascular diseases, like detected strokes, myocardial infarctions, revascularization procedures, arrythmias (eg atrial fibrillation).

OTHER OUTCOMES:
Treatment compliance and secondary treatment targets | 15 years
  Secondary endpoints include significant cardiovascular diseases, like detected strokes, myocardial infarctions, revascularization procedures, and arrhythmia (e.g. atrial fibrillation). Treatment compliance is monitored based on drug purchases and achieving clinically set secondary prevention targets (e.g., cholesterol levels, blood pressure, and blood glucose levels).

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital Tampere Heart Centre, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be only shared according to European General Data Protection Regulation (GDPR) and other regulation as appropriate.